CLINICAL TRIAL: NCT03850431
Title: Using Behavioral Economics to Enhance Appointment Reminders and Reduce Missed Visits
Acronym: No Show
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Iowa City VA Health Care System (U.S. Federal Agency); VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 17-134; HX002449 (Other Grant/Funding Number: VA Health Services Research and Development)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-10

CONDITIONS: Appointment Reminders
Keywords: Behavioral Economics; Mental Health; Veterans; Veterans Health; Primary Care; Appointments and Schedules
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The primary objective is to systematically develop and test the effectiveness of a series of changes to appointment letters in a cluster RCT with the goal of reducing no-shows and increasing access. First, the investigators will iteratively obtain feedback and refine messages in draft interventions (Aim 1). Then evaluate the effects of four enhanced appointment reminder interventions informed by BE and the Theory of Planned Behavior, and compare them to usual care and each other (Aims 2 and 3). Appointments will be randomly allocated to one of the four interventions or usual care at the provider-level, with providers blinded to allocation. The trial will be conducted at eight locations across VAPORHCS in both mental health and primary care. The investigators will also conduct a qualitative assessment with key informants (Aim 4) to provide data that will be useful for future implementation (if intervention is effective) or suggest modifications to the intervention (if ineffective).
Masking Description: The intervention arms were assigned letters and the statistician was blinded for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Social Norms + Behavioral Instructions (Experimental): Clinics assigned a letter with two types of nudges (Social Norms + Behavioral Instructions)
  Interventions: Behavioral: Social Norms + Behavioral Instructions
- Caring + Consequences for Others + Behavioral Instructions (Experimental): Clinics assigned a letter with three types of nudges (Caring + Consequences for Others + Behavioral Instructions)
  Interventions: Behavioral: Caring + Consequences for Others + Behavioral Instructions
- Caring + Consequences for Self + Behavioral Instructions (Experimental): Clinics assigned a letter with three types of nudges (Caring + Consequences for Self + Behavioral Instructions)
  Interventions: Behavioral: Caring + Consequences for Self + Behavioral Instructions
- Combination of all Nudges (Experimental): Clinics assigned a letter with a combination of all types of nudges (Behavioral: Caring + Consequences for Others + Consequences for Self + Social Norms + Behavioral Instructions)
  Interventions: Behavioral: Caring + Consequences for Others + Consequences for Self + Social Norms + Behavioral Instructions
- Usual Care (No Intervention): Clinics assigned to usual care. Usual care consisted of a letter with basic appointment information on date, location, and phone number(s) for scheduling changes

INTERVENTIONS:
Behavioral: Social Norms + Behavioral Instructions — A letter with two types of nudges. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
  Arms: Social Norms + Behavioral Instructions
Behavioral: Caring + Consequences for Others + Behavioral Instructions — A letter with three types of nudges. One suggests that the institution cares about the patient. One highlights a potential negative consequence for others if the patient no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
  Arms: Caring + Consequences for Others + Behavioral Instructions
Behavioral: Caring + Consequences for Self + Behavioral Instructions — A letter with three types of nudges. One suggests that the institution cares about the patients. One highlights potential negative consequences for the patient if s/he no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
  Arms: Caring + Consequences for Self + Behavioral Instructions
Behavioral: Caring + Consequences for Others + Consequences for Self + Social Norms + Behavioral Instructions — A letter with all types of nudges combined. One suggests that the institution cares about the patients. One highlights a potential negative consequence for others if the patient no-shows. One highlights potential negative consequences for the patient if s/he no-shows. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
  Arms: Combination of all Nudges

SUMMARY:
"No-shows," or missed visits are a persistent problem in all health care systems. They contribute to worsened patient access, longer wait times, and inefficient use limited health care resources. The VA's no-show rate has shown no improvement in years, resulting in a staggering 9 million ambulatory no-shows in Fiscal Year (FY) 2015. Appointment reminders are an essential and proven element to addressing no-shows but major research gaps exist. Behavioral economics (BE) and allied fields offer key insights that are relevant to developing innovation in the field of appointment reminders. Adding "nudges" informed by concepts such as social norms, behavioral intentions, clear instructions, and potential negative consequences to the Veteran and others is a novel but evidence-based way to create enhanced appointment reminders. Seemingly small changes to appointment letters can create measurable shifts in appointment attendance and no-shows. Even more, these behavioral nudges can produce large benefits when taken to scale and compounded across a population.

This project will address several aims, including: developing BE-informed messages to incorporate into enhanced appointment reminders; evaluating the effect of several versions of enhanced appointment reminders; and identifying potential barriers and facilitators to widespread implementation of enhanced appointment reminder messages.

DETAILED DESCRIPTION:
Objectives: The overarching objective of this proposal is to test the effectiveness of simple and scalable enhancements to appointment reminders in reducing no-shows, and prepare for larger-scale implementation.

Plan: "No-shows," or missed visits are a persistent problem in all health care systems. They contribute to worsened patient access, longer wait times, and inefficient use limited health care resources. The VA's no-show rate has shown no improvement in years, resulting in a staggering 9 million ambulatory no-shows in FY2015. Appointment reminders are an essential and proven element to addressing no-shows but major research gaps exist. Behavioral economics (BE) and allied fields offer key insights that are relevant to developing innovation in the field of appointment reminders. Adding "nudges" informed by concepts such as social norms, behavioral intentions, clear instructions, and potential negative consequences to the Veteran and others is a novel but evidence-based way to create enhanced appointment reminders. Seemingly small changes to appointment letters can create measurable shifts in appointment attendance and no-shows. Even more, these behavioral nudges can produce large benefits when taken to scale and compounded across a population.

The investigators will address the following aims:

1. Aim 1: Develop and iteratively refine BE-informed messages based on Veterans' perceptions, and incorporate them into enhanced appointment reminders.
2. Aim 2: Determine the effect of four versions of enhanced appointment reminders on measures relevant to treatment access, compared with usual reminders.
3. Aim 3: Evaluate differences in treatment effect associated with four versions of enhanced appointment reminders.
4. Aim 4: Characterize potential barriers and facilitators to widespread implementation of enhanced appointment reminder messages.

Methods: The investigators will first determine the validity of a series of draft messages, which are informed by concepts and principles from BE, psychology, and related fields and will be included in the intervention; the investigators will also explore potential mechanisms of action, and measure any harms by assessing Veterans' perceptions of the messages (Aim 1). After intervention refinement, the investigators will conduct a cluster randomized controlled trial to test 4 interventions, consisting of variations in nudges included in appointment letters, and compare them to usual appointment letters (Aims 2 and 3). The trial will be conducted at VA Portland Health Care System (VAPORHCS) in primary care and mental health clinics. The investigators will evaluate changes in no-show rates, attendance and cancellation rates and appointment wait times. Finally, the investigators will conduct a qualitative assessment with key informants to inform potential barriers and facilitators to implementation of revised appointment reminders (Aim 4).

Relevance to VA's Mission: This proposal directly addresses two of the six Health Services Research and Development Service (HSR&D) priority areas: access and mental and behavioral health. First, reducing no-shows is likely to improve efficiency of access to care and reduce wait time. Second, this proposal includes a focus on interventions in mental health settings, which have especially high no-show rates and may have more potential for improvement.

Medical Subject Heading Terms: Economics, Behavioral; Mental Health; Healthcare Quality, Access, and Evaluation

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be a minimum of 18 years old.
* All subjects will be patients with scheduled outpatient appointments (either primary care or mental health) in the VA Portland Health Care System.
* Race and ethnicity will not be used in determining inclusion or exclusion of subjects.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34516 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan R. Teo, MD MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teo AR, Metcalf EE, Strange W, Call AA, Tuepker A, Dobscha SK, Kaboli PJ. Enhancing Usability of Appointment Reminders: Qualitative Interviews of Patients Receiving Care in the Veterans Health Administration. J Gen Intern Med. 2021 Jan;36(1):121-128. doi: 10.1007/s11606-020-06183-5. Epub 2020 Sep 9. PMID 32909229
- [Result] Zikmund-Fisher BJ, Tuepker A, Metcalf EE, Strange W, Teo AR. Applying user-centered design in the development of nudges for a pragmatic trial to reduce no-shows among veterans. Patient Educ Couns. 2022 Jun;105(6):1620-1627. doi: 10.1016/j.pec.2021.10.024. Epub 2021 Oct 23. PMID 34756639
- [Result] Lafferty M, Strange W, Kaboli P, Tuepker A, Teo AR. Patient Sense of Belonging in the Veterans Health Administration: A Qualitative Study of Appointment Attendance and Patient Engagement. Med Care. 2022 Sep 1;60(9):726-732. doi: 10.1097/MLR.0000000000001749. Epub 2022 Jul 26. PMID 35880766
- [Result] Teo AR, Niederhausen M, Handley R, Metcalf EE, Call AA, Jacob RL, Zikmund-Fisher BJ, Dobscha SK, Kaboli PJ. Using Nudges to Reduce Missed Appointments in Primary Care and Mental Health: a Pragmatic Trial. J Gen Intern Med. 2023 Jul;38(Suppl 3):894-904. doi: 10.1007/s11606-023-08131-5. Epub 2023 Jun 20. PMID 37340264

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Primary Care Appointments: Usual Care: A Primary Care appointment letter that includes basic appointment information on date, location, and phone number(s) for scheduling changes.
- Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions: A Primary Care appointment letter with three types of nudges. One suggests that the institution cares about the patients. One highlights potential negative consequences for the patient if s/he no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions: A Primary Care appointment letter with three types of nudges. One suggests that the institution cares about the patient. One highlights a potential negative consequence for others if the patient no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Primary Care Appointments: Social Norms + Behavioral Instructions: A Primary Care appointment letter with two types of nudges. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Primary Care Appointments: Combination of All Nudges: A Primary Care appointment letter with all types of nudges combined. One suggests that the institution cares about the patients. One highlights a potential negative consequence for others if the patient no-shows. One highlights potential negative consequences for the patient if s/he no-shows. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Mental Health Appointments: Usual Care: A Mental Health appointment letter that includes basic appointment information on date, location, and phone number(s) for scheduling changes.
- Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions: A Mental Health appointment letter with three types of nudges. One suggests that the institution cares about the patients. One highlights potential negative consequences for the patient if s/he no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions: A Mental Health appointment letter with three types of nudges. One suggests that the institution cares about the patient. One highlights a potential negative consequence for others if the patient no-shows. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Mental Health Appointments: Social Norms + Behavioral Instructions: A Mental Health appointment letter with two types of nudges. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
- Mental Health Appointments: Combination of All Nudges: A Mental Health appointment letter with all types of nudges combined. One suggests that the institution cares about the patients. One highlights a potential negative consequence for others if the patient no-shows. One highlights potential negative consequences for the patient if s/he no-shows. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
Period: Overall Study
Arm/Group | Primary Care Appointments: Usual Care | Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions | Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions | Primary Care Appointments: Social Norms + Behavioral Instructions | Primary Care Appointments: Combination of All Nudges | Mental Health Appointments: Usual Care | Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions | Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions | Mental Health Appointments: Social Norms + Behavioral Instructions | Mental Health Appointments: Combination of All Nudges
Started (Some patients had appointments in multiple arms of the study, so the sum of participants in each arm will not equal the number of unique participants in the trial.) | 10929; 50 Clinics | 13465; 51 Clinics | 13525; 50 Clinics | 9223; 52 Clinics | 12556; 51 Clinics | 3737; 51 Clinics | 3996; 44 Clinics | 4844; 48 Clinics | 4760; 46 Clinics | 3354; 45 Clinics
Completed (Some patients had appointments in multiple arms of the study, so the sum of participants in each arm will not equal the number of unique participants in the trial.) | 5584; 47 Clinics | 7287; 48 Clinics | 6196; 43 Clinics | 5056; 44 Clinics | 6543; 49 Clinics | 2184; 46 Clinics | 2167; 39 Clinics | 2863; 45 Clinics | 2860; 43 Clinics | 2142; 42 Clinics
Not Completed | 5345; 3 Clinics | 6178; 3 Clinics | 7329; 7 Clinics | 4167; 8 Clinics | 6013; 2 Clinics | 1553; 5 Clinics | 1829; 5 Clinics | 1981; 3 Clinics | 1900; 3 Clinics | 1212; 3 Clinics

BASELINE CHARACTERISTICS:
Population: Some participants had appointments with clinics that were randomized to different arms. In this table, participants are only counted once within the 5 primary care arms and once within the 5 mental health arms, according to their first primary care or mental health appointment. This table's total column includes the 4014 participants who had appointments in both primary care and mental health twice - once in each. Summary statistics for age & gender are based on the 32,946 unique participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Appointments: Usual Care | Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions | Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions | Primary Care Appointments: Social Norms + Behavioral Instructions | Primary Care Appointments: Combination of All Nudges | Mental Health Appointments: Usual Care | Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions | Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions | Mental Health Appointments: Social Norms + Behavioral Instructions | Mental Health Appointments: Combination of All Nudges | Total
Number analyzed (Participants) | 4916 | 6592 | 5759 | 4353 | 5920 | 1641 | 1666 | 2305 | 2250 | 1558 | 36960
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall number of participants includes 4014 participants who had appointments in both primary care and mental health in the total twice. Summary statistics for age are based on the 32,946 unique participants.
  years
    Primary Care: number analyzed (Participants) | 4916 | 6592 | 5759 | 4353 | 5920 | 0 | 0 | 0 | 0 | 0 | 27540
    Primary Care | 65.60 (14.44) | 64.81 (14.85) | 62.77 (15.92) | 62.87 (16.08) | 62.62 (16.14) |  |  |  |  |  | 63.75 (15.53)
    Mental Health: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1641 | 1666 | 2305 | 2250 | 1558 | 9420
    Mental Health |  |  |  |  |  | 50.06 (15.95) | 49.49 (16.22) | 51.39 (16.16) | 49.37 (15.85) | 49.29 (15.75) | 49.99 (16.01)
Sex/Gender, Customized [Number; unit: participants] — Self-identified gender according to medical record Population: The overall number of participants includes 4014 participants who had appointments in both primary care and mental health in the total twice. Summary statistics for gender are based on the 32,946 unique participants.
  participants
    Primary Care - Female: number analyzed (Participants) | 4916 | 6592 | 5759 | 4353 | 5920 | 0 | 0 | 0 | 0 | 0 | 27540
    Primary Care - Female | 349 | 564 | 839 | 444 | 587 |  |  |  |  |  | 2738
    Primary Care - Male: number analyzed (Participants) | 4916 | 6592 | 5759 | 4353 | 5920 | 0 | 0 | 0 | 0 | 0 | 27540
    Primary Care - Male | 4567 | 6028 | 4920 | 3909 | 5333 |  |  |  |  |  | 24757
    Mental Health - Female: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1641 | 1666 | 2305 | 2250 | 1558 | 9420
    Mental Health - Female |  |  |  |  |  | 300 | 403 | 477 | 362 | 306 | 1848
    Mental Health - Male: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1641 | 1666 | 2305 | 2250 | 1558 | 9420
    Mental Health - Male |  |  |  |  |  | 1341 | 1263 | 1828 | 1888 | 1252 | 7572
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall includes both primary care and mental health counts together.
  Participants
    Primary Care: number analyzed (Participants) | 4916 | 6592 | 5759 | 4353 | 5920 | 0 | 0 | 0 | 0 | 0 | 27540
    Primary Care: American Indian or Alaska Native | 65 | 91 | 71 | 58 | 72 |  |  |  |  |  | 357
    Primary Care: Asian | 49 | 60 | 45 | 70 | 57 |  |  |  |  |  | 281
    Primary Care: Native Hawaiian or Other Pacific Islander | 37 | 46 | 39 | 45 | 63 |  |  |  |  |  | 230
    Primary Care: Black or African American | 155 | 218 | 172 | 147 | 199 |  |  |  |  |  | 891
    Primary Care: White | 3888 | 5340 | 4540 | 3488 | 4760 |  |  |  |  |  | 22016
    Primary Care: More than one race | 61 | 70 | 59 | 54 | 63 |  |  |  |  |  | 307
    Primary Care: Unknown or Not Reported | 661 | 767 | 833 | 491 | 706 |  |  |  |  |  | 3458
    Mental Health: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1641 | 1666 | 2305 | 2250 | 1558 | 9420
    Mental Health: American Indian or Alaska Native |  |  |  |  |  | 19 | 25 | 37 | 37 | 29 | 147
    Mental Health: Asian |  |  |  |  |  | 27 | 21 | 33 | 34 | 25 | 140
    Mental Health: Native Hawaiian or Other Pacific Islander |  |  |  |  |  | 12 | 12 | 29 | 25 | 20 | 98
    Mental Health: Black or African American |  |  |  |  |  | 83 | 69 | 96 | 101 | 87 | 436
    Mental Health: White |  |  |  |  |  | 1251 | 1289 | 1823 | 1730 | 1147 | 7240
    Mental Health: More than one race |  |  |  |  |  | 33 | 30 | 42 | 47 | 36 | 188
    Mental Health: Unknown or Not Reported |  |  |  |  |  | 216 | 220 | 245 | 276 | 214 | 1171

OUTCOME MEASURES:

1. Primary Outcome: No-Show Rate
Description: The percentage of total appointments that are classified as a no-show, relative to the total number of appointments scheduled. The numerator ("no-shows") consists of appointments marked as a no-show and appointments canceled by the patient or clinic after the appointment time. The denominator ("total appointments") consists of no-shows and completed appointments. For calculation of missed appointments, canceled appointments are not included in the number of units analyzed. The numerator is multiplied by 100 to arrive at a percentage.
Time Frame: 1 year
Population: The number of participants analyzed is greater than listed in Participant Flow because these results include two additional arms listed for analysis: all 4 Primary Care intervention arms, and all 4 Mental Health intervention arms. These were not individual arms to which participants were randomized but rather a combination of arms for purposes of analysis.
  The number of appointments analyzed is greater than the number of participants because some participants had multiple appointments.
Measure: Number; unit: percentage of appointments no showed
Units Other Than Participants: Appointment
Groups:
- Primary Care - All 4 Primary Care Intervention Arms Combined: Combination of all 4 Primary Care intervention arms. Note: this was not an individual study arm to which participants were randomized, but rather a combination of arms for purposes of data analysis.
- Mental Health - All 4 Mental Health Intervention Arms Combined: Combination of all 4 Mental Health intervention arms. Note: this was not an individual study arm to which participants were randomized, but rather a combination of arms for purposes of data analysis.
Arm/Group | Primary Care Appointments: Usual Care | Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions | Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions | Primary Care Appointments: Social Norms + Behavioral Instructions | Primary Care Appointments: Combination of All Nudges | Primary Care - All 4 Primary Care Intervention Arms Combined | Mental Health Appointments: Usual Care | Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions | Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions | Mental Health Appointments: Social Norms + Behavioral Instructions | Mental Health Appointments: Combination of All Nudges | Mental Health - All 4 Mental Health Intervention Arms Combined
Number analyzed (Participants) | 5584 | 7287 | 6196 | 5056 | 6543 | 22624 | 2184 | 2167 | 2863 | 2860 | 2142 | 7779
Number analyzed (Appointment) | 9721 | 12321 | 7492 | 7688 | 8889 | 36390 | 6144 | 5750 | 8131 | 8411 | 6984 | 29276
percentage of appointments no showed | 11.9 | 11.1 | 10.5 | 12.1 | 10.6 | 11.1 | 18.0 | 19.2 | 21.9 | 20.0 | 18.9 | 20.1
Statistical Analysis 1: Comparison: Primary Care Appointments: Usual Care vs Primary Care - All 4 Primary Care Intervention Arms Combined; Test type: Other; p = 0.145, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.139, 95% CI 2-sided [0.956 to 1.357]
Statistical Analysis 2: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions; Test type: Other; p = 0.298, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.912 to 1.35]
Statistical Analysis 3: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions; Test type: Other; p = 0.127, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.178, 95% CI 2-sided [0.955 to 1.452]
Statistical Analysis 4: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Combination of All Nudges; Test type: Other; p = 0.286, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.117, 95% CI 2-sided [0.911 to 1.37]
Statistical Analysis 5: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Social Norms + Behavioral Instructions; Test type: Other; p = 0.183, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.925 to 1.504]
Statistical Analysis 6: Comparison: Mental Health Appointments: Usual Care vs Mental Health - All 4 Mental Health Intervention Arms Combined; Test type: Other; p = 0.209, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.903 to 1.595]
Statistical Analysis 7: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions; Test type: Other; p = 0.463, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.144, 95% CI 2-sided [0.799 to 1.638]
Statistical Analysis 8: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions; Test type: Other; p = 0.074, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.331, 95% CI 2-sided [0.972 to 1.822]
Statistical Analysis 9: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Combination of All Nudges; Test type: Other; p = 0.306, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.169, 95% CI 2-sided [0.867 to 1.577]
Statistical Analysis 10: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Social Norms + Behavioral Instructions; Test type: Other; p = 0.373, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.845 to 1.565]

2. Secondary Outcome: Cancellation Rate
Description: The percentage of scheduled appointments that are marked as canceled.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of appointments cancelled
Units Other Than Participants: Appointments
Groups:
- Mental Health Appointments: Combination of All Nudges: A Mental Health appointment letter with all four types of nudges combined. One suggests that the institution cares about the patients. One highlights a potential negative consequence for others if the patient no-shows. One highlights potential negative consequences for the patient if s/he no-shows. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
Arm/Group | Primary Care Appointments: Usual Care | Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions | Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions | Primary Care Appointments: Social Norms + Behavioral Instructions | Primary Care Appointments: Combination of All Nudges | Primary Care - All 4 Primary Care Intervention Arms Combined | Mental Health Appointments: Usual Care | Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions | Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions | Mental Health Appointments: Social Norms + Behavioral Instructions | Mental Health Appointments: Combination of All Nudges | Mental Health - All 4 Mental Health Intervention Arms Combined
Number analyzed (Participants) | 5584 | 7287 | 6196 | 5056 | 6543 | 22624 | 2184 | 2167 | 2863 | 2860 | 2142 | 7779
Number analyzed (Appointments) | 10339 | 13070 | 8223 | 8251 | 9715 | 39259 | 6843 | 6343 | 8841 | 9270 | 7648 | 32012
percentage of appointments cancelled | 6.0 | 5.7 | 8.9 | 6.8 | 8.5 | 7.3 | 10.2 | 9.3 | 8.0 | 9.3 | 8.7 | 8.8
Statistical Analysis 1: Comparison: Primary Care Appointments: Usual Care vs Primary Care - All 4 Primary Care Intervention Arms Combined; Test type: Other; p = 0.153, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.923, 95% CI 2-sided [0.826 to 1.03]
Statistical Analysis 2: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Caring + Consequences for Self + Behavioral Instructions; Test type: Other; p = 0.252, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.911, 95% CI 2-sided [0.777 to 1.068]
Statistical Analysis 3: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Caring + Consequences for Others + Behavioral Instructions; Test type: Other; p = 0.413, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.941, 95% CI 2-sided [0.815 to 1.088]
Statistical Analysis 4: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Combination of All Nudges; Test type: Other; p = 0.41, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.946, 95% CI 2-sided [0.83 to 1.079]
Statistical Analysis 5: Comparison: Primary Care Appointments: Usual Care vs Primary Care Appointments: Social Norms + Behavioral Instructions; Test type: Other; p = 0.11, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.887, 95% CI 2-sided [0.766 to 1.027]
Statistical Analysis 6: Comparison: Mental Health Appointments: Usual Care vs Mental Health - All 4 Mental Health Intervention Arms Combined; Test type: Other; p = 0.14, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.833, 95% CI 2-sided [0.654 to 1.062]
Statistical Analysis 7: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Caring + Consequences for Self + Behavioral Instructions; Test type: Other; p = 0.404, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.882, 95% CI 2-sided [0.657 to 1.184]
Statistical Analysis 8: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Caring + Consequences for Others + Behavioral Instructions; Test type: Other; p = 0.072, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.743, 95% CI 2-sided [0.538 to 1.027]
Statistical Analysis 9: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Combination of All Nudges; Test type: Other; p = 0.057, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.778, 95% CI 2-sided [0.6 to 1.008]
Statistical Analysis 10: Comparison: Mental Health Appointments: Usual Care vs Mental Health Appointments: Social Norms + Behavioral Instructions; Test type: Other; p = 0.637, Regression, Logistic; Logistic regression with clustering for clinics and patients; Odds Ratio (OR) = 0.932, 95% CI 2-sided [0.697 to 1.247]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for one year.
Description: Participants were not individually enrolled in this study, and there was no direct contact with participants. For this reason we were not able to monitor mortality. We monitored for other potential adverse events and protocol deviations. One adverse event occurred, for which we were able to determine the intervention but not whether it was regarding a primary care or a mental health appointment. To allow for accurate reporting, primary care and mental health arms were combined by intervention.
Groups:
- Usual Care: An appointment reminder that includes basic appointment information on date, location, and phone number(s) for scheduling changes.
- Combination of All Nudges: A letter with all types of nudges combined. One suggests that the institution cares about the patients. One highlights a potential negative consequence for others if the patient no-shows. One highlights potential negative consequences for the patient if s/he no-shows. One points out the common behavior of attending appointments. And one provides clear, specific instructions for making appointment changes. The appointment reminder also includes usual care (basic appointment information on date, location, and phone number(s) for scheduling changes).
Arm/Group | Usual Care | Caring + Consequences for Self + Behavioral Instructions | Caring + Consequences for Others + Behavioral Instructions | Social Norms + Behavioral Instructions | Combination of All Nudges
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7768 | 0/9454 | 0/9059 | 0/7196 | 0/8685
Other Adverse Events (participants affected / at risk) | 0/7768 | 0/9454 | 0/9059 | 1/7196 | 0/8685
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=7768) | Caring + Consequences for Self + Behavioral Instructions (N=9454) | Caring + Consequences for Others + Behavioral Instructions (N=9059) | Social Norms + Behavioral Instructions (N=7196) | Combination of All Nudges (N=8685)
Emotional distress (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Veteran called patient advocate stating that content of the Social Norms letter was offensive and not appropriate in addressing why the Veteran missed an appointment. Identifiable participant information was unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03850431/Prot_SAP_000.pdf